CLINICAL TRIAL: NCT06443515
Title: Evaluation of Respiratory Trends During Blood Transfusions in Newborns.
Brief Title: Respiratory Trends During Blood Transfusions in Newborns.
Acronym: ARTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6438
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Blood Transfusion Complication; Blood Transfusion Associated Adverse Reactions; Respiratory Complication; Respiratory Morbidity
MeSH Terms: conditions — Transfusion Reaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Other): All infants undergoing blood transfusions will be enrolled in the study
  Interventions: Diagnostic Test: lung ultrasound

INTERVENTIONS:
Diagnostic Test: lung ultrasound — Lung ultrasound examinations will be performed within 6 hours before and after blood transfusion to assess interstitial-alveolar fluid retention and calculate a LUS score

SUMMARY:
The prevalence of transfusion reactions is between 1 and 11% of transfusions. Most reactions are mild and do not pose a life-threatening risk to the patient. More serious problems may be the only manifestations that lead to suspicion of a transfusion reaction.

Most noninfectious transfusion reactions are immune-mediated. Two main types of reactions can be distinguished: TACO (transfusion associated cardiac overload, which is a cardiogenic pulmonary edema) and TRALI (transfusion related acute lung injury, non-cardiogenic pulmonary edema).

Although TRALI are diagnoses of exclusion, the presence of noncardiogenic pulmonary edema and respiratory problems in the vicinity of blood product transfusions should raise suspicion. Other signs of TRALI are hypotension and tachycardia, while in TACO arterial hypertension with positive water balance can be observed.

According to previous reports, the prevalence of transfusion reactions in the neonatal population is approximately 8%. Factors associated with these reactions are low birth weight and low gestational age. However, diagnostic criteria of respiratory transfusion reactions are not uniform across studies, and often the generic terms "acute lung injury" have been used.

Therefore, the primary objective of this study is to evaluate the respiratory trend during blood transfusions; secondary objectives are the study of risk factors for the development of respiratory worsening and the possible association with complications.

ELIGIBILITY:
Inclusion Criteria:

* admitted newborns requiring blood transfusions as per local practice and/or international guidelines

Exclusion Criteria:

* newborns with major malformations
* need for palliative care
* lack of informed consent

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Changes in lung ultrasound score (LUS score) before and after transfusions | within 6 hours before and after the transfusion
  LUS score according to previous publications (Brat et al., 2015) will be calculated
Changes in non-invasive peripheral oxygen saturation/fraction of inspired oxygen (SFR) before and after transfusions | within 6 hours before and after the transfusion
  non-invasive peripheral oxygen saturation/fraction of inspired oxygen (SFR) will be calculated from clinical charts: data validated by caregivers (primary nurses) will be extracted from the electronic charts to calculate this ratio

SECONDARY OUTCOMES:
Changes in ventilatory parameters (mean airway pressure) for patients on nasal continuous positive airway pressure (nCPAP) or mechanical ventilation | within 6 hours before and after the transfusion
  MAP as displayed by ventilators will be recorded as median values

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Nobile, MD, PhD, MSc, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No